CLINICAL TRIAL: NCT00773981
Title: Transrectal Vacuum Assisted Drainage: A NEW METHOD OF TREATING ANASTOMOTIC LEAKAGE AFTER RECTAL RESECTION. A Prospective Randomized Multicenter Study in Cooperation With "The Danish Colorectal Cancer Group"
Brief Title: Transrectal Vacuum Assisted Drainage: A New Method of Treating Anastomotic Leakage After Rectal Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Braun Aesculap (Unknown)
Responsible Party: Dr Carl Frederik Nagell, Hamlet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-B-2007-061
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-10

CONDITIONS: Colorectal Surgery
Keywords: anastomotic leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Endoluminal vacuum therapy.
  Interventions: Procedure: Transrectal vacuum assisted drainage
- 2 (No Intervention): Patients not receiving vacuum therapy should be treated with a catheter with daily rinsing for a minimum of 7 days.

INTERVENTIONS:
Procedure: Transrectal vacuum assisted drainage — Treatment with vacuum drainage (VD) is a new method primarily developed for wound therapy. The principle of the method is application of negative pressure on the wound surface with the help of a sponge that is connected to a pump. Sponge dressings should be changed 3 times pr week as long as vacuum therapy is used. If there has been no development of granulation tissue or no shrinking of the cavity in 3 weeks Vacuum therapy can be stopped. Maximum vacuum therapy is 8 weeks.
  Arms: 1

SUMMARY:
Anastomotic leakage is a major and potentially mortal complication with an incidence of 10-13% after resection of the rectum. For patients showing no clinical signs of peritonitis, the traditional method has been a conservative treatment with transrectal rinsing. This treatment is often associated with a very protracted postoperative course with healing times of up to a year or more for the anastomotic leakage.

Treatment with vacuum drainage (VD) is a new method primarily developed for wound therapy.

The objective of this study is to investigate the effects of transrectal vacuum treatment on the healing of anastomotic leakage after rectum resection in a prospective, randomized, controlled multicentre trial in 60 patients found to develop clinically significant anastomotic leakages after elective rectal resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically significant* anastomotic leakage after intended curative rectal resection (LAR) for rectal cancer with primary anastomosis.
* Patients whose operation did not include ileostomy must have surgery to create a stoma within two days after beginning of the vacuum therapy and before randomization. Anastomotic leakage must have been diagnosed within 21 days of the primary operation.
* Patients with and without preoperative radiation therapy may participate.
* Groups will be formed accordingly, because patients who had preoperative radiation therapy heal more slowly.
* Patients with anastomotic leakage (diagnosed by endoscopic or radiology techniques) and clinical signs and symptoms indicating a health impairment (fever, pain, elevated creatinine levels).
* Anastomotic leakage after rectal cancer surgery

Exclusion Criteria:

* Informed consent
* Age < 18 years
* Acute surgery
* Leakage diagnosed more than 21 days after the primary operation
* Patient does not consent to temporary ileostomy
* Anastomosis technically inaccessible for vacuum-assisted drainage
* Small intestine visible in abscess cavity
* Residual cancer tissue in the pelvic cavity
* Suspicion of fistulation between the abscess cavity and internal genitalia, urinary tract system, or small intestines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Healing time of the anastomotic leakage | 1 year

SECONDARY OUTCOMES:
Salvage surgery (abdominal reoperation with debridement of anastomosis) | 1 month
Duration of fever and antibiotic treatment | 2 months
Duration of hospital stay | 2 monts
Number of visits in the outpatient clinic / number of sponge changes | 8 weeks
Functional result, defined as +/- closure of temporary ileostomy | 2 years
Functional result evaluated by examination of the anal physiology in a smaller patient population (supplementary trial protocol) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl F Nagell, MD, Principal Investigator — Hamlet Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Hvidovre, Denmark